CLINICAL TRIAL: NCT04828226
Title: Clonidine to Prevent Postictal Delirium After ElectroConvulsive Therapy: a Randomised, Placebo-controlled, Triple-blind, Single-centre Trial.
Brief Title: Clonidine to Prevent Delirium After Electroconvulsive Therapy.
Acronym: ECaTa
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BECD-3-21
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder; Catatonia; Bipolar Disorder; Delirium Postseizure
Keywords: Electroconvulsive Therapy; ECT; Clonidine; Postictal Delirium; Postseizure Delirium; Postictal Agitation; Postseizure Agitation; CAM-ICU; RASS
MeSH Terms: conditions — Depressive Disorder, Major; Catatonia; Bipolar Disorder | interventions — Clonidine; calcium D-pantothenate, L-cysteine drug combination

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomised, placebo-controlled, triple blind, single-centre, two-arm parallel groups superiority trial assessing incidence and severity of postictal delirium.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After randomisation in RedCap, a study nurse otherwise not involved in the trial will store group allocation in an envelope (labelled with the patients study identifier, name and date of birth) in a closed cupboard accessible to the post-anaesthesia care team member preparing the study drug, but not the treating or assessing team. After a patient's trial completion, the envelope and its content will be destroyed.
  Therefore, the treating team, the patient as well as the data collecting personnel is blinded to group allocation. The bottles containing study drug or placebo are identical and are identically labelled with "Study Drug" and the patients name by the independent post-anaesthesia care member preparing the study drug before ECT sessions start. Data analysts will be blinded as well because allocation to verum or placebo is only known to the study nurse randomising patients and preparing the envelopes needed for drug preparation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The study drug (clonidine 2 mcg/kg) is diluted in 100 ml sodium chloride 0.9 % by trained post-anaesthesia care staff not involved in the study.
  At admission, electrocardiogram, non-invasive blood pressure and pulse oximetry is installed, a peripheral venous line established and supplemental oxygen applied.
  The study drug will be given intravenously over 10 minutes at least 10 minutes before induction of anaesthesia.
  Electroconvulsive therapy will be conducted according to hospital standard (Etomidate 0.2 mg/kg, Suxamethonium 1.0 mg/kg, isolated limb technique, THYMATRON® SYSTEM IV, Somatics Inc., Lake Bluf, Illinois, USA) adjusted to the patient's condition. Seizure quality will be assessed, prolonged seizure activity terminated with propofol 0.2 - 0.3 mg/kg. Severe agitation (Richmond Agitation and Sedation Score (RASS) > 1) needing intervention will be treated with propofol or lorazepam. Patients will be assessed for delirium using CAM-ICU at 20 minutes after induction.
  Interventions: Drug: Clonidine
- Control (Placebo Comparator): The placebo will be created by diluting 1ml of sodium chloride 0.9% in 100ml of sodium chloride in a sterile manner prior to application. The container will be identically labelled as the verum. The placebo will be applied by the same team members named above via the same route (intravenously), with the same speed and the same timing. All other parts of the procedure are identical as to the procedure described above.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine — Clonidine 2mcg/kg Body Weight diluted in 100ml sodium chloride 0.9% compared to placebo (sodium chloride 0.9% alone) given over 10 minutes, 10 minutes prior to electroconvulsive therapy.
  Other Names: Verum
  Arms: Intervention
Drug: Placebo — Sodium chloride 0.9% 100ml given over 10minutes, 10 minutes prior to electroconvulsive therapy.
  Arms: Control

SUMMARY:
Electroconvulsive therapy (ECT) is a highly effective treatment for some psychiatric disorders like major depressive or bipolar disorder, but may lead to agitation and delirium after the procedure in up to 65% of patients. This can have negative side effects and be dangerous for patient and attending staff. Clonidine, a central-acting alpha2-receptor agonist, is an approved antihypertensive medication with known sedative side effects. Clonidine's newer but more expensive successor, dexmedetomidine, has recently shown its potential to reduce this kind of delirium. The investigators therefore hypothesise that pre-treatment with 2 mcg/kg clonidine prior to electroconvulsive therapy will significantly reduce the incidence of postictal delirium. This potentially makes a highly efficient treatment for patients with otherwise refractory psychiatric illness safer and more accessible.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is a highly efficacious therapy for psychiatric disorders, especially major depressive disorder, bipolar disorder and catatonia resistant to psychopharmacology or drug-psychotherapy combination therapy. At therapy induction, usually a series of 10-12 ECT sessions is planned with two to three days in between sessions. Thereafter, maintenance therapy can be continued with longer session intervals thereafter to avoid relapses and to support further drug and psychotherapy treatment. Without maintenance therapy, relapses can happen in up to 80% of all patients within one year.

Nowadays conducted under general anaesthesia (etomidate in the investigator's centre) and muscle relaxation (suxamethonium) to prevent adverse events, ECT can be challenging for the anaesthesiologist, as it usually leads to rapid cardiovascular changes such as sudden bradycardia due to vagal discharge, followed by sympathetic counter regulation associated with tachycardia and hypertension. For the patient, known immediate side effects are headache in about 30% and postictal confusion and delirium in up to 65%. This confusional state can lead to involuntary movements and agitation and therefore be harmful for patients and attending staff. It usually resolves within 45 minutes but nevertheless seems to be linked with adverse side effects like persistent retrograde amnesia. Identified risk factors are long seizure time and pre-existing catatonic features. Postictal delirium has been classified by Kikuchi et. al. into four categories from no delirium, mild, moderate or severe delirium. Moderate to severe delirium needing restraints or sedative medication like benzodiazepines or Propofol was present 36% of patients, which is in line with older data. The more severe forms of delirium are easily recognised in clinical practice because of the need for intervention. When including mild forms, delirium was present in 52% of all patients in the study of Kikuchi et al. In newer studies using a more sensitive tool (CAM-ICU, Confusion Assessment Method - Intensive Care Unit) to assess the presence of delirium, the rates are up to 65% at 10 minutes after ECT stimulation respectively 10 minutes after arrival in the post-anaesthesia care unit. CAM-ICU is a brief but sensitive test, which has been extensively validated in the intensive care setting. Therefore, it seems that postictal delirium is frequently underdiagnosed in clinical practice. As we know from the intensive care literature, even hypoactive forms of delirium are associated with higher complication rates and higher mortality and therefore cannot be neglected.

In previous small studies, premedication with promethazine, midazolam and dexmedetomidine successfully reduced incidence of postictal delirium. Dexmedetomidine, a highly selective, relatively short acting alpha2-agonist, has been more extensively studied in the setting of ECT and has recently been able to show his potency to reduce postictal delirium by a third when given as a bolus pre-induction in a randomised controlled trial.

In this prospective, randomised, placebo-controlled, triple-blind, single-centre, two-arm parallel groups superiority trial, the investigators aim to lower incidence and severity of postictal delirium and agitation using a pre-induction dose of 2 mcg/kg clonidine intravenously compared to placebo (sodium chloride). The investigators also hypothesise, that a pre-induction dose of clonidine will reduce incidence of postictal agitation, the need for sedative rescue medication and the need for short-acting antihypertensive medication. It therefore might increase patient safety and cost effectiveness without prolonging post-anaesthesia care unit stay or negatively affecting treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and more;
* Scheduled for an elective series of ambulatory ECT sessions at the University Hospital Bern;
* Informed Consent as documented by signature (Appendix Informed Consent Form).

Exclusion Criteria:

* Contraindications to the study drug, e. g. known allergy or hypersensitivity, hypotension, bradycardia, higher grade atrioventricular block;
* On regular Clonidine for another indication (e.g. arterial hypertension)
* Patients undergoing emergency ECT;
* Unable to consent (incapable of judgment, next-of-kin consent necessary or under tutelage);
* Inability to follow the procedures of the study, e. g. due to language barrier;
* Previous enrolment into the current study;
* Participation in another study with investigational drug within the 30 days preceding and during the present study;
* Enrolment of the investigator, his/her family members, employees and other dependent persons.
* Women who are pregnant or breast feeding;
* Intention to become pregnant during the course of the study;
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration (and 4 weeks thereafter), such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases. Female participants who are surgically sterilised / hysterectomised or post-menopausal for longer than 2 years are not considered as being of child bearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2021-04-27 (Actual); Primary Completion 2026-07-27 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delirium after electroconvulsive therapy over all (twelve) ECT sessions | 20 minutes after muscle relaxation
  The primary outcome is delirium after electroconvulsive therapy over all (twelve) ECT sessions. The presence of delirium will be assessed using Confusion Assessment Method - Intensive Care Unit (CAM-ICU). To be able to perform the test correctly, the patient must be awake enough. This will be assessed using the Richmond-Agitation-Sedation-Scale (RASS) first ranging from -5 (unarousable) to +4 (combative)

SECONDARY OUTCOMES:
Incidence of mild agitation | post-anaesthesia care unit stay (up to 2 hours)
  RASS +1, needing verbal command or short restraint < 1 minute
Incidence of severe agitation | post-anaesthesia care unit stay (up to 2 hours)
  RASS > 1, needing restraint > 1 minute or rescue medication)
Use of rescue medication | post-anaesthesia care unit stay (up to 2 hours)
  medication, dose, route
Duration of seizure activity | during procedure (estimated to be on average 10-15 minutes)
  seconds
Quality of seizure activity | during procedure (estimated to be on average 10-15 minutes)
  ideal, sufficient, insufficient
Seizure Quality Index | during procedure (estimated to be on average 10-15 minutes)
  Seizure Quality Index (Kranaster et al., Eur Arch Psychiatry Clin Neurosci 2018) ranging from 0 to 5. Higher index indicates better response to treatment.
Need for seizure terminating medication | during procedure (estimated to be on average 10-15 minutes)
  medication, dose, route
Total number of electroconvulsive therapy sessions | whole treatment course (12 ECT sessions, about 4 weeks)
  number
Reason for terminating or continuing the electroconvulsive series | whole treatment course (12 ECT sessions, about 4 weeks)
  failure, response, remission, other reason
Length of post-anaesthesia care unit stay | post-anaesthesia care unit stay (up to 2 hours)
  minutes
Incidence of desaturation | post-anaesthesia care unit stay (up to 2 hours)
  Oxygen saturation by pulse oximetry < 75%, irrespective of duration
Incidence of hypotension | during procedure (estimated to be on average 10-15 minutes)
  any measurement with mean arterial pressure < 55 mmHg
Incidence of bradycardia | post-anaesthesia care unit stay (up to 2 hours)
  heart rate < 50 bpm for more than 1 minute
Cardiovascular changes needing intervention | post-anaesthesia care unit stay (up to 2 hours)
  number and type
Use of cardiovascular medication | post-anaesthesia care unit stay (up to 2 hours)
  medication, dose, route
Adverse events potentially attributable to ECT | whole treatment course (12 ECT sessions, about 4 weeks)
  diagnosis
Adverse events potentially attributable to Study Drug | whole treatment course (12 ECT sessions, about 4 weeks)
  diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wüthrich, Prof, MD, Principal Investigator — Department of Anaesthesiology and Pain Medicine, Bern University Hospital, University of Bern
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Bern University Hospital, University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No